CLINICAL TRIAL: NCT02401802
Title: Low-fiber Diet for Colorectal Cancer Screening Colonoscopy. Randomized Clinical Trial. Dietcol Study
Brief Title: Low-fiber Diet for Colorectal Cancer Screening Colonoscopy
Acronym: DIETCOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Marco Antonio Alvarez Gonzalez, MD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DIETCOL
Record Dates: First submitted 2015-03-17; First posted 2015-03-30 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Colonic Diseases
Keywords: Colonoscopy; Diet; Polyethylene glycols; Efficacy; Personal satisfaction; Colorectal cancer screening
MeSH Terms: conditions — Colonic Diseases; Personal Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-residue diet (Experimental): The experimental group will receive 4 days of low-residue diet Laxative 4 liters polyethylene glycol 4000 in split fashion.
  Interventions: Dietary Supplement: Low-residue diet
- Usual care (Active Comparator): The control group will receive 3 days of low-residue diet followed by 24 hours of liquid diet.
  Laxative 4 liters polyethylene glycol 4000 in split fashion.
  Interventions: Dietary Supplement: Usual care

INTERVENTIONS:
Dietary Supplement: Low-residue diet — Subjects will be instructed by members of the research team to follow a standardized low residue diet for 4 days
  Arms: Low-residue diet
Dietary Supplement: Usual care — Subjects will be instructed by members of the research team to follow a low-residue diet for 3 days followed by 24 hours of liquid diet
  Arms: Usual care

SUMMARY:
This trial will compare the efficacy of 2 different sets of dietary recommendations to be followed before colon cleansing for colorectal cancer screening colonoscopy.

DETAILED DESCRIPTION:
There is no enough evidence in the literature to recommend a low-fiber diet for screening colonoscopy. Although evidence of benefit of a liquid diet is minimal and there is a growing body of evidence about the benefits of a liberalized diet, a high degree of heterogeneity in the clinical trials comparing the diet modifications before colonoscopy prevents a formal recommendation in current guidelines. A low-fiber diet the day before colonoscopy may result in same efficacy of bowel cleanliness, with an improved tolerability and acceptability.

All consecutive patients of a population-based colorectal screening cancer program referred for a colonoscopy will be invited to participate in the study. After obtaining informed consent, they will be randomized to one of the groups: liquid diet or low-fiber diet. The will be interviewed by a registered research nurse, and they will be provided with written instructions for bowel preparation and questionnaires for registering the data of the study. The day of the colonoscopy, questionnaires will be collected and endoscopists blinded for the study bowel preparation will perform the colonoscopy. Patients will be contacted for adverse events and a general satisfaction questionnaire, 3 days after colonoscopy.

ELIGIBILITY:
Inclusion criteria:

* Consecutive patients referred for a colonoscopy in a population-based colorectal screening program.

Exclusion criteria:

* Unwillingness to participate.
* Inability to follow instructions
* Active inflammatory bowel disease
* Incomplete colonoscopies for technical reasons or contraindication as evaluated by the endoscopist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Inadequate bowel preparation. | 1 hour after the colonoscopy
  The efficacy of bowel preparation will be rated by blinded endoscopists using the Boston Bowel Preparation Scale (BBPS). Colonoscopies with a BBPS score of less than 5 points, or any segment rated less than 2 points will be considered with an inadequate bowel preparation

SECONDARY OUTCOMES:
Cecal intubation rate | 1 hour after the colonoscopy
  Ratio of successful cecal intubations in each study arm
Adenoma detection rate | 1 hour after the colonoscopy
  Ratio of polyps and adenomas detected in each study arm
Polyp detection rate | 1 hour after the colonoscopy
  Ratio of polyps and adenomas detected in each study arm
Abdominal pain | 6 hours after finishing bowel preparation
  Each participant will rate his/her experience in an analogue visual scale
Nausea | 6 hours after finishing bowel preparation
  Each participant will rate his/her experience in an analogue visual scale
Hunger | 6 hours after finishing bowel preparation
  Each participant will rate his/her experience in an analogue visual scale
Bloating | 6 hours after finishing bowel preparation
  Each participant will rate his/her experience in an analogue visual scale
Adverse events | 30 days after the colonoscopy
  Description of all spontaneously reported adverse events.
Adherence to the planned bowel cleansing method (questionnaire) | 6 hours after finishing bowel preparation
  Each participant will rate his/her experience in a questionnaire.
Acceptability of the preparation (interference with work, leisure activities or sleep | 6 hours after finishing bowel preparation
  Each participant will rate his/her experience in a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Antonio Alvarez González, MD, PhD, Principal Investigator — Parc de Salut Mar
Locations (1):
- Hospital del Mar, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Soweid AM, Kobeissy AA, Jamali FR, El-Tarchichi M, Skoury A, Abdul-Baki H, El-Zahabi L, El-Sayyed A, Barada KA, Sharara AI, Mourad F, Arabi A. A randomized single-blind trial of standard diet versus fiber-free diet with polyethylene glycol electrolyte solution for colonoscopy preparation. Endoscopy. 2010 Aug;42(8):633-8. doi: 10.1055/s-0029-1244236. Epub 2010 Jul 9. PMID 20623443
- [Derived] Alvarez-Gonzalez MA, Pantaleon MA, Flores-Le Roux JA, Zaffalon D, Amoros J, Bessa X, Seoane A, Pedro-Botet J; PROCOLON group. Randomized Clinical Trial: A Normocaloric Low-Fiber Diet the Day Before Colonoscopy Is the Most Effective Approach to Bowel Preparation in Colorectal Cancer Screening Colonoscopy. Dis Colon Rectum. 2019 Apr;62(4):491-497. doi: 10.1097/DCR.0000000000001305. PMID 30844973